CLINICAL TRIAL: NCT02298309
Title: Test and Treat TB: A Proof of Concept Trial in South Africa
Acronym: Siyasiza
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); AIDS Healthcare Foundation (Other)
Responsible Party: Principal Investigator, Ingrid V. Bassett, MD, MPH, Associate Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2014P001173/MGH; R21AI110264 (NIH)
Record Dates: First submitted 2014-11-18; First posted 2014-11-21 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Tuberculosis
Keywords: TB; HIV; Test and Treat; Linkage
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention): Patients in the usual care arm will be screened for tuberculosis (TB) on a mobile unit and referred for treatment according to the current standard of care in South Africa
- Test-and-Treat Intervention (Active Comparator): Patients in the intervention arm will partake in a Test-and-Treat TB strategy involving mobile GeneXpert MTB/RIF testing, facilitated TB treatment initiation, SMS reminders for clinic visits, and cashless incentives.
  Interventions: Other: Test-and-Treat TB

INTERVENTIONS:
Other: Test-and-Treat TB
  Arms: Test-and-Treat Intervention

SUMMARY:
The purpose of this study is (1) to establish the feasibility, yield, and clinical impact of a "Test & Treat TB" strategy on a mobile HIV screening unit in South Africa and (2) to assess the cost and cost-effectiveness of this mobile, integrated HIV/TB screening strategy for maximizing linkage to TB care and treatment completion.

ELIGIBILITY:
Inclusion Criteria:

* English or Zulu speaking
* presenting for screening at mobile unit
* voluntarily undergoing HIV testing
* able and willing to give informed consent
* willing to share HIV and TB test results
* willing to attend one of six local clinics for treatment
* access to a mobile phone

Exclusion Criteria:

* pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4815 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Number of patients who complete tuberculosis treatment | 6 months

SECONDARY OUTCOMES:
Proportion of mobile testers screened for tuberculosis | 20 months
Proportion of eligible participants able to produce sputum samples | 20 months
Prevalence of TB among those tested | 20 months
Prevalence of tuberculosis and rifampin resistance | 20 months
  The GeneXpert test can detect rifampin resistant strains of tuberculosis
Distribution of TB symptoms ascertained from TB symptom screen questionnaire | 20 months
Proportion returning to the mobile tester for TB test result | 20 months
Linkage to TB care (first visit to a local TB treatment site ascertained from clinic record) | 1 month
ART initiation date as documented by clinic record for those HIV co-infected | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid V Bassett, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- iThembalabantu Clinic/AIDS Healthcare Foundation, Durban, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bassett IV, Forman LS, Govere S, Thulare H, Frank SC, Mhlongo B, Losina E. Test and Treat TB: a pilot trial of GeneXpert MTB/RIF screening on a mobile HIV testing unit in South Africa. BMC Infect Dis. 2019 Feb 4;19(1):110. doi: 10.1186/s12879-019-3738-4. PMID 30717693

DOCUMENTS (1):
  • Study Protocol (2017-05-26): https://cdn.clinicaltrials.gov/large-docs/09/NCT02298309/Prot_000.pdf